CLINICAL TRIAL: NCT02229877
Title: A Study in Healthy Subjects to Assess the Effect of Intragastric pH and Fasting on the Multiple-Dose Pharmacokinetics of AF-219
Brief Title: A Study to Assess the Effect of Intragastric pH and Fasting on the Pharmacokinetics of Gefapixant (AF-219/MK-7264)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 7264-011; AF219-011 (Other: Afferent Pharmaceuticals)
Record Dates: First submitted 2014-08-27; First posted 2014-09-03 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Omeprazole; Gefapixant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gefapixant + Omeprazole (Experimental): Gefapixant oral tablets (25mg, 50 mg, 150 mg) administered twice daily for 18 days
  + Omeprazole oral capsules (40 mg) administered twice daily for 8.5 days
  Interventions: Drug: Omeprazole; Drug: Gefapixant

INTERVENTIONS:
Drug: Omeprazole — 40 mg oral capsules administered twice daily for 8.5 days
  Other Names: Prilosec
Drug: Gefapixant — Gefapixant oral tablet (25 mg administered as a divided 50 mg tablet) administered twice daily for 2 days
  Other Names: AF-219; MK-7264
Drug: Gefapixant — Gefapixant oral tablet (50 mg tablet) administered twice daily for 8 days
  Other Names: AF-219; MK-7264
Drug: Gefapixant — Gefapixant oral tablet (150 mg administered as three 50 mg tablets) administered twice daily for 8 days
  Other Names: AF-219; MK-7264

SUMMARY:
The purpose of this study is to: determine the effect of stomach pH on the multiple dose pharmacokinetics (PK) of gefapixant (AF-219); assess the effect of multiple doses of gefapixant on various sensory assessments; and, assess the safety and tolerability of gefapixant.

ELIGIBILITY:
Inclusion Criteria:

Must be informed of the nature of the study and have provided written informed voluntary consent;

Able to speak, read, and understand English;

Healthy males or females, of any race, between 18 and 55 years of age, inclusive;

Body mass index (BMI) >18.5 and <32.0 kg/m2 and weigh 50 - 100 kg;

In good general health ;

Non-smokers for at least 5 years;

If a female of child-bearing potential (i.e., have not undergone a hysterectomy or bilateral oophorectomy) or not post-menopausal (defined as no menses for at least 12 months), agree to use 2 forms of acceptable birth control; or if a male, they and/or their partner of child-bearing potential agree to use 2 forms of acceptable birth control;

Exclusion Criteria:

Any disease or condition that might affect drug absorption, metabolism, or excretion or clinically significant cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, gastrointestinal, immunological, dermatological, neurological, or psychiatric disease;

Clinically significant illness or clinically significant surgery within 4 weeks before the administration of study medication;

Any past sinus surgery, upper respiratory tract infection within 2 weeks before dosing, or history of hay fever during the time of the year that dosing will be taking place;

History of GERD, heartburn, or nausea more than once a month, or any similar symptoms requiring the regular use of antacids, or any use of H2 histamine blockers or proton pump inhibitors within 12 months of Screening;

Have a positive screening test for Helicobacter pylori;

QTcB >450 msec in males or >460 msec in females;

Known or suspected hypersensitivity or allergic reaction to any of the components of gefapixant or omeprazole capsules;

If female, is pregnant or breast feeding, or has a positive pregnancy test pre dose;

Blood loss or blood donation of >550 mL within 90 days or plasma donation >500 mL within 14 days before administration of the first dose of study drug;

Chronic use of any systemic medications; use of a drug therapy known to induce or inhibit hepatic drug metabolism within 30 days before the first dose of study medication; or use of any medications including antacids, high dose multivitamins, nutritional supplements, and herbal preparations, within 14 days before the first dose of study drug;

Past or current history or evidence of drug or alcohol abuse, use of any recreational soft drugs (e.g., marijuana) within 3 months of screening, use of any hard drugs (such as cocaine, phencyclidine (PCP), and crack) within 1 year of screening, and/or a positive screen for substances of abuse or alcohol at screening or pre dose;

Ingestion of grapefruit or grapefruit juice within 48 hours before dose administration;

Positive urine cotinine test at Screening or Day 1 pre dose;

Positive screen for hepatitis B surface antigen (HBsAg), hepatitis C antibody, or human immunodeficiency virus (HIV) antibody;

Receipt of an investigational product or device, or participation in a drug research study within a period of 30 days (or 5 half lives of the drug, whichever is longer) before the first dose of study medication;

Receipt of an investigational immunomodulator or monoclonal antibody within 180 days (or 5 half lives, whichever is longer) before the first dose of study medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2015-05-22 (Actual)

PRIMARY OUTCOMES:
Effect of Intragastric pH on gefapixant PK | At pre-dose (time 0) and at 1, 2, 3, 5, 8, and 12 hours post dose
  Analysis of variance (ANOVA) will be performed on log normal-transformed Cmax and AUC0-t values to determine the extent of a drug interaction, if any, of omeprazole on the plasma gefapixant PK parameters. These analyses will be conducted for both fed and fasted conditions and the 50 mg and 150 mg treatments.

SECONDARY OUTCOMES:
Effect of Fasting on gefapixant PK | At pre-dose (time 0) and at 1, 2, 3, 5, 8, and 12 hours post dose
  ANOVA will be performed on log normal-transformed Cmax and AUC0-t values to determine if fasting affects plasma gefapixant PK parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Terry O'Reilly, M.D., Principal Investigator — Celerion

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Gupta P, Hussain A, Ford AP, Smith S, Nussbaum JC, Stoch A, Iwamoto M. Clinical Formulation Bridging of Gefapixant, a P2X3-Receptor Antagonist, for the Treatment of Chronic Cough. Clin Pharmacol Drug Dev. 2022 Sep;11(9):1054-1067. doi: 10.1002/cpdd.1105. Epub 2022 May 5. PMID 35510785